CLINICAL TRIAL: NCT06390150
Title: Midline Versus Dorsolateral Spinal Cord Stimulation for Post-surgical Neuropathic Pain (MIDL-SCS Trial)
Brief Title: Midline Versus Dorsolateral Spinal Cord Stimulation for Post-surgical Neuropathic Pain
Acronym: MIDL-SCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Lutz Weise, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MIDL-SCS
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Pain, Postoperative; Neuropathic Pain
Keywords: Spinal cord stimulation; Post intra-thoracic surgery pain syndrome
MeSH Terms: conditions — Pain, Postoperative; Neuralgia

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a placebo-controlled, crossover, randomized clinical trial of the intervention dorsolateral spinal cord stimulation (DL-SCS) for the indication post-surgical focal neuropathic pain. Study arm order will be randomly generated and known only to the programmer. Once participants have crossed over into all study arms, they will be set on their best program and enter long-term observation.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- DL-SCS Only (Experimental): The DL-SCS electrode will be activated with a high-frequency paresthesia-free program.
  Interventions: Device: Spinal Cord Stimulator
- Stimulation Off (Placebo Comparator): Both electrodes will be programmed for sham stimulation.
  Interventions: Device: Spinal Cord Stimulator
- M-SCS Only (Experimental): The M-SCS electrode will be activated with a high-frequency, paresthesia free program.
  Interventions: Device: Spinal Cord Stimulator
- DL-SCS + M-SCS (Experimental): Both DL-SCS and M-SCS will be activated with high-frequency, paresthesia free programs.
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — The spinal cord stimulator is an implantable pulse generator connected to electrodes with leads that stimulate the spinal cord. The device is programmed to deliver therapeutic stimulation to treat pain.

SUMMARY:
The goal of this interventional study is to learn if dorsolateral spinal cord stimulation (DL-SCS) can treat focal post-surgical, medically refractory neuropathic pain. The main question it aims to answer is:

- How does DL-SCS compare to traditional SCS and no treatment for treating post-surgical neuropathic pain?

Participants will be asked to

* trial combinations of stimulation across blocks of weeks (randomized cross-over)
* rate their pain after each stimulation trial

DETAILED DESCRIPTION:
Neuropathic pain resulting from injury to the somatosensory nervous system can be a persistent and debilitating condition of spontaneous and unprovoked symptoms. For patients with chronic neuropathic pain that does not respond to conservative therapy, spinal cord stimulation (SCS) may be considered. SCS has been established as an effective and sustained treatment for neuropathic pain, but may deliver treatment to more than just the pain area. Dorsolateral spinal cord stimulation (DL-SCS) may provide a more focal alternate target for spinal stimulation. The aim of this study is to investigate DL-SCS as a therapeutic option for post-surgical, medically refractory neuropathic pain. This is a prospective, randomized, double-blind controlled crossover trial to investigate the efficacy of DL-SCS and midline SCS (M-SCS) compared to sham stimulation for the diagnosis of post-surgical neuropathic pain. Each participant will be implanted with two electrodes and will crossover into each stimulation program in a randomized order to serve as their own control.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of neuropathic pain following a surgical procedure
2. A minimum of 50% of pain should be limited to one body part, defined as one limb or one side of trunk.
3. Failed conservative therapies (medication, physiotherapy)
4. Disability more than 6 months

Exclusion criteria

1. Previous implantation with SCS (i.e. revision surgery)
2. Any underlying condition that would preclude an MRI
3. Untreated psychiatric conditions or substance use disorder
4. Existing medical conditions that would preclude from SCS (history of recurrent infections, uncontrolled cancer, etc.)
5. Surgically treatable lesion (e.g. spinal stenosis, disc herniation)
6. Lack of capacity (e.g. significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Numerical Rating Scale (NRS) for pain intensity | Baseline and at 4, 6, 8, 10, 52, 104 weeks post-surgery
  The primary outcome is the self-reported difference in change from baseline of the severity of pain quantified in the Numerical Rating Scale. This will be assessed at baseline (pre-surgery) and at regular follow-up appointments.

SECONDARY OUTCOMES:
Change in score on Oswestry Disability Index | Baseline and at 4, 6, 8, 10, 52, 104 weeks post-surgery
  Assesses a patient's quality of life in relation to back pain on a 10-section questionnaire. A low score indicates no disability and a high score indicates severe disability.
Change in score on EuroQol 5 Dimension Questionnaire | Baseline and at 4, 6, 8, 10, 52, 104 weeks post-surgery
  Assesses overall quality of life in five dimensions including mobility, self-care, daily routine, pain, and anxiety/depression. A low score indicates poor health and a high score indicates excellent health.
Change in morphine equivalents used | Baseline and at 4, 6, 8, 10, 52, 104 weeks post-surgery
  Measures patient pain by assessing the amount of pain medication taken by a patient. Higher usage indicates a greater level of pain and a lower usage indicates a lower level of pain.
Change in score on the Brief Pain Inventory Short Form | Baseline and at 4, 6, 8, 10, 52, 104 weeks post-surgery
  Assesses the impact of pain on a patient's quality of life. A high score indicates a severe impact and a lower score indicates minimal impact.
Change in score on the 12-item Short Form Survey | Baseline and at 4, 6, 8, 10, 52, 104 weeks post-surgery
  Assesses how a patient's health impacts their quality of life. A higher score indicates a better quality of life, and a low score indicates a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Weise, MD, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth Health Science Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No